CLINICAL TRIAL: NCT04350866
Title: Enhancing Access to Insomnia (EASI) Care: Implementing Brief Behavioral Treatment for Insomnia in Primary Care Mental Health Integration Clinics
Brief Title: Enhancing Access to Insomnia (EASI) Care in VA PCMHI Clinics
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Pittsburgh Healthcare System (U.S. Federal Agency); VA Maryland Health Care System (U.S. Federal Agency); Durham VA Health Care System (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IIR 19-340
Record Dates: First submitted 2020-03-31; First posted 2020-04-17 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Insomnia
Keywords: Veterans; stepped-wedge design; hybrid implementation-effectiveness trial; primary care mental health integration
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Minneapolis VAMC: BBTI; ERIC strategies
  Interventions: Behavioral: Expert Recommendations for Implementing Change bundle of strategies; Behavioral: Brief Behavioral Treatment for Insomnia
- Philadelphia VAMC: BBTI; ERIC strategies
  Interventions: Behavioral: Expert Recommendations for Implementing Change bundle of strategies; Behavioral: Brief Behavioral Treatment for Insomnia
- Durham VAMC: BBTI; ERIC strategies
  Interventions: Behavioral: Expert Recommendations for Implementing Change bundle of strategies; Behavioral: Brief Behavioral Treatment for Insomnia
- Baltimore VAMC: BBTI; ERIC strategies
  Interventions: Behavioral: Expert Recommendations for Implementing Change bundle of strategies; Behavioral: Brief Behavioral Treatment for Insomnia

INTERVENTIONS:
Behavioral: Expert Recommendations for Implementing Change bundle of strategies — * Develop a formal implementation blueprint/checklist
  * Conduct educational meetings
  * Develop and distribute educational materials
  * Organize implementation meetings
  * Facilitation
  * Increase demand with marketing to patients
  * Promote adaptability
  Other Names: ERIC
Behavioral: Brief Behavioral Treatment for Insomnia — An adapted version of Cognitive Behavioral Therapy for Insomnia (CBT-I) that is focused on behavioral components stimulus control and sleep restriction (the four rules):
  1. Reduce time awake in bed.
  2. Don't go to bed unless ready for sleep.
  3. Don't stay in bed unless asleep.
  4. Get up and out of bed at the same time everyday.
  Delivered weekly to bi-weekly over 4-6 sessions, with each session typically 30 minutes or less, consistent with other interventions delivered in PCMHI.
  Other Names: BBTI

SUMMARY:
This multi-site project (four VA Medical Centers) will test two approaches to improving the delivery of a behavioral insomnia treatment in the Primary Care setting to Veterans. The first approach is training providers to deliver Brief Behavioral Treatment for Insomnia (BBTI). The second approach is to give providers trained in BBTI additional support and resources to enhance their ability to deliver BBTI, what we call implementation. This project will measure delivery of BBTI over four phases: (1) pre-training; (2) pre-implementation; (3) implementation; and (4) post-implementation.

The main questions to answer:

Does delivery of BBTI improve with training alone and does it improve further with the addition of implementation support?

Does delivery of BBTI remain at similar levels after implementation support is removed?

Do Veterans who engage in BBTI reduce their insomnia symptoms?

DETAILED DESCRIPTION:
Chronic insomnia, one of the most common health problems among Veterans, significantly impacts health, function, and quality of life. Cognitive Behavioral Therapy for Insomnia (CBTI) is the first line treatment; however, despite efforts to train VA clinicians to deliver CBTI, there are still significant barriers to providing adequate access to insomnia care. Up to 44% of Veterans seen in Primary Care report insomnia, making it an optimal clinical setting for improving access to insomnia care. Furthermore, Brief Behavioral Treatment for Insomnia (BBTI), adapted from CBTI as a briefer, more flexible treatment, is easily delivered by Primary Care Mental Health Integration (PCMHI) clinicians and can greatly improve access to care for Veterans with insomnia. Yet, simply training PCMHI clinicians to deliver BBTI is not enough. Implementation strategies are needed for successful uptake, adoption, and sustainable delivery of care.

This stepped-wedge, hybrid III implementation-effectiveness trial involves four VA Medical Centers: Baltimore, Durham, Minneapolis, and Philadelphia. The hybrid design allows for testing of implementation and treatment effectiveness. The stepped-wedge design allows for fewer sites to achieve adequate power as all sites are exposed to BBTI training (BBTI) and BBTI + Implementation Strategies (BBTI+IS). The target sample are PCMHI clinicians and the impact of a bundle of strategies on the success of sustainable delivery of BBTI in Primary Care. Retrospective data collected from VA electronic health records will be used to obtain variables of interest related to Veteran treatment outcomes and data related to PCMHI clinician delivery of BBTI.

We will compare the impact PCMHI clinicians trained to deliver BBTI vs. the impact of BBTI training plus 12-months of access to an implementation strategy bundle (BBTI+IS). BBTI+IS vs. BBTI training alone is expected to result in more Veterans with access to insomnia care in PCMHI. We will also compare delivery of BBTI across all four phases, from pre-training to post-implementation. We will also measure Veteran-level outcomes for insomnia severity and PCMHI clinician fidelity on delivery of BBTI.

Outcome measures have been updated to reflect study protocol and analyses more accurately. Some of the prespecified Primary and Secondary Outcome Measures have been combined with one removed due to no data collection. The results reported reflect data that has been collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

All Veterans in Primary Care and Primary Care Mental Health Integration (PCMHI) at the participating sites.

Exclusion Criteria:

Not meeting above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four (4) VAMCs will be randomized to the order in which they will receive the intervention (stepped wedge). At each VAMC, retrospective data will be collected on Veterans who receive care in Primary Care and Primary Care Mental Health Integration (PCMHI). Our goal is to identify Veterans who engage in Brief Behavioral Treatment for Insomnia (BBTI) in a PCMHI clinic. Our goal is to collect data on at least 332 Veterans during the implementation phase (n=83 Veterans/site).
Sampling Method: Non-Probability Sample
Enrollment: 277920 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam D. Bramoweth, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bramoweth AD, Hough CE, O'Brien EM, Klingaman EA, Deininger CJ, Ulmer CS, Boudreaux-Kelly MY, McCoy JL, Youk AO. Implementing brief behavioral treatment for insomnia in Department of Veterans Affairs Primary Care Mental Health Integration clinics: Reach outcomes from a hybrid type 3 effectiveness-implementation trial. Psychol Serv. 2025 Aug;22(3):409-422. doi: 10.1037/ser0000924. Epub 2025 Jan 2. PMID 39745672
- See also: Brief Behavioral Treatment for Insomnia (BBTI introduction for patients and providers) — https://www.youtube.com/watch?v=ZhFS5MLKrv0
- See also: The 2 Processes that Regulate Sleep and the 4 Rules to Improve Your Sleep — https://www.youtube.com/watch?v=WmxphTTAg6U

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four (4) VA Medical Centers (VAMC) were enrolled in this project. Within each VAMC, we identified Veterans (Participants) who engaged in care within PCMHI clinics. Veterans' data was collected retrospectively starting from January 1, 2020 until July 31, 2024. PCMHI providers (Staff) at each site were also consented for feedback and intervention fidelity ratings. 277,920 unique Veteran Participants and Staff were enrolled across all phases; however, enrollment differs at each phase.
Pre-assignment Details: Staff did not participate in the Pre-Training phase. Data collection for a site could have ranged from 36 to 54 months (including phases 1-4; excluding the 1-month BBTI training period January 1, 2021 - January 31, 2021).
Groups:
- Minneapolis VAMC: All sites underwent a 12-month pre-training period (phase 1) before undergoing training (month 0) for BBTI. Then sites were randomized to 0, 6, 12, or 18 months of the Pre-Implementation (phase 2), followed by 12 months of Implementation (phase 3, ERIC strategies were accessible and supported during this phase), and 12 months of Post-Implementation monitoring (phase 4).
  *This site was assigned to: Pre-Training, then Implementation (Month 1-12), then Post-Implementation (Month 13-24). Note, this site was randomized to skip Pre-Implementation (phase 2).
- Philadelphia VAMC: All sites underwent a 12-month pre-training period (phase 1) before undergoing training (month 0) for BBTI. Then sites were randomized to 0, 6, 12, or 18 months of the Pre-Implementation (phase 2), followed by 12 months of Implementation (phase 3, ERIC strategies were accessible and supported during this phase), and 12 months of Post-Implementation monitoring (phase 4).
  *This site was assigned to: Pre-Training, then Pre-Implementation (Month 1-6), Implementation (Month 7-18), then Post-Implementation (Month 19-30).
- Durham VAMC: All sites underwent a 12-month pre-training period (phase 1) before undergoing training (month 0) for BBTI. Then sites were randomized to 0, 6, 12, or 18 months of the Pre-Implementation (phase 2), followed by 12 months of Implementation (phase 3, ERIC strategies were accessible and supported during this phase), and 12 months of Post-Implementation monitoring (phase 4).
  *This site was assigned to: Pre-Training, then Pre-Implementation (Month 1-12), Implementation (Month 13-24), then Post-Implementation (Month 25-36).
- Baltimore VAMC: All sites underwent a 12-month pre-training period (phase 1) before undergoing training (month 0) for BBTI. Then sites were randomized to 0, 6, 12, or 18 months of the Pre-Implementation (phase 2), followed by 12 months of Implementation (phase 3, ERIC strategies were accessible and supported during this phase), and 12 months of Post-Implementation monitoring (phase 4).
  *This site was assigned to: Pre-Training, then Pre-Implementation (Month 1-18), Implementation (Month 19-30), then Post-Implementation (Month 31-42).
Period: Pre-Training (12 Months)
Arm/Group | Minneapolis VAMC | Philadelphia VAMC | Durham VAMC | Baltimore VAMC
Started (Number of participants in each phase (period) will not match as this is the number of patients, from the electronic medical records, that are engaging in care at each site within each phase (period).) | 74207 | 42663 | 56179 | 42218
PCMHI Participants | 4725 | 4481 | 3939 | 2833
Primary Care Participants | 69482 | 38182 | 52240 | 39385
Staff | 0 | 0 | 0 | 0
Completed | 74207 | 42663 | 56179 | 42218
Not Completed | 0 | 0 | 0 | 0
Period: Pre-Implementation (0, 6, 12, 18 Months)
Arm/Group | Minneapolis VAMC | Philadelphia VAMC | Durham VAMC | Baltimore VAMC
Started (Number of participants in each phase (period) will not match as this is the number of patients, from the electronic medical records, that are engaging in care at each site within each phase (period).) | 0 (This site did not go through this phase.) | 30888 (Month 1-6) | 56655 (Month 1-12) | 42568 (Month 1-18)
PCMHI Participants | 0 | 2759 | 4792 | 3580
Primary Care Participants | 0 | 28124 | 51858 | 38979
Staff | 0 | 5 | 5 | 9
Completed | 0 | 30888 | 56655 | 42568
Not Completed | 0 | 0 | 0 | 0
Period: Implementation (12 Months)
Arm/Group | Minneapolis VAMC | Philadelphia VAMC | Durham VAMC | Baltimore VAMC
Started (*This phase (period) used for Baseline data. Number of participants in each phase (period) will not match as this is the number of patients, from the electronic medical records, that are engaging in care at each site within each phase (period).) | 75154 (Month 1-12) | 37582 (Month 7-18) | 49859 (Month 13-24) | 33558 (Month 19-30)
PCMHI Participants | 4924 | 3927 | 2975 | 2258
Primary Care Participants | 70223 | 33650 | 46878 | 31291
Staff | 7 | 5 | 6 | 9
Completed | 75154 | 37582 | 49859 | 33558
Not Completed | 0 | 0 | 0 | 0
Period: Post-Implementation (12 Months)
Arm/Group | Minneapolis VAMC | Philadelphia VAMC | Durham VAMC | Baltimore VAMC
Started (Number of participants in each phase (period) will not match as this is the number of patients, from the electronic medical records, that are engaging in care at each site within each phase (period).) | 65411 (Month 13-24) | 33401 (Month 19-30) | 46797 (Month 25-36) | 32677 (Month 31-42)
PCMHI Participants | 3669 | 3107 | 2511 | 2324
Primary Care Participants | 61735 | 30289 | 44280 | 30344
Staff | 7 | 5 | 6 | 9
Completed | 65411 | 33401 | 46797 | 32677
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants from all sites identified in the Implementation phase in PCMHI and Primary Care, and Staff from all sites identified among all phases.
Groups:
- Minneapolis VAMC: All sites underwent a 12-month pre-training period (phase 1) before undergoing training (month 0) for BBTI. Then sites were randomized to 0, 6, 12, or 18 months of the Pre-Implementation (phase 2), followed by 12 months of Implementation (phase 3, ERIC strategies were accessible and supported during this phase), and 12 months of Post-Implementation monitoring (phase 4).
  *This site was assigned to: Pre-Training, then Implementation (Month 1 - Month 12), then Post-Implementation (Month 13-24). Note, this site was randomized to skip Pre-Implementation (phase 2).
- Staff: Staff consented from all 4 sites in the Pre-Implementation, Implementation, and Post-Implementation phases.
- Total: Total of all reporting groups
Arm/Group | Minneapolis VAMC | Philadelphia VAMC | Durham VAMC | Baltimore VAMC | Staff | Total
Number analyzed (Participants) | 75147 | 37577 | 49853 | 33549 | 27 | 196153
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants from all sites identified in the Implementation phase in PCMHI and Primary Care, and Staff from all sites identified among all phases. Population: Veteran and Staff participants analyzed separately
  years
    PCMHI Participants: number analyzed (Participants) | 4924 | 3927 | 2975 | 2258 | 0 | 14084
    PCMHI Participants | 57.18 (17.57) | 55.35 (16.05) | 52.75 (15.23) | 54.19 (14.35) |  | 55.25 (16.26)
    Primary Care Participants: number analyzed (Participants) | 70223 | 33650 | 46878 | 31291 | 0 | 182042
    Primary Care Participants | 65.46 (15.87) | 64.08 (15.70) | 60.57 (15.16) | 61.69 (14.90) |  | 63.30 (15.63)
    Staff: number analyzed (Participants) | 0 | 0 | 0 | 0 | 27 | 27
    Staff |  |  |  |  | 40.23 (9.50) | 40.23 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants] — Participants from all sites identified in the Implementation phase in PCMHI and Primary Care, and Staff from all sites identified among all phases. Population: Veteran and Staff participants analyzed separately
  Participants
    PCMHI Participants: number analyzed (Participants) | 4924 | 3927 | 2975 | 2258 | 0 | 14084
    PCMHI Participants: Female | 832 | 646 | 557 | 561 |  | 2596
    PCMHI Participants: Male | 4092 | 3281 | 2418 | 1697 |  | 11488
    Primary Care Participants: number analyzed (Participants) | 70223 | 33650 | 46878 | 31291 | 0 | 182042
    Primary Care Participants: Female | 4610 | 3167 | 5936 | 4386 |  | 18099
    Primary Care Participants: Male | 65613 | 30483 | 40942 | 26905 |  | 163943
    Staff: number analyzed (Participants) | 0 | 0 | 0 | 0 | 27 | 27
    Staff: Female |  |  |  |  | 22 | 22
    Staff: Male |  |  |  |  | 5 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants from all sites identified in the Implementation phase in PCMHI and Primary Care, and Staff from all sites identified among all phases. Population: Veteran and Staff participants analyzed separately
  Participants
    PCMHI Participants: number analyzed (Participants) | 4924 | 3927 | 2975 | 2258 | 0 | 14084
    PCMHI Participants: White | 4024 | 1679 | 1276 | 784 |  | 7763
    PCMHI Participants: Non-White | 495 | 1985 | 1543 | 1345 |  | 5368
    PCMHI Participants: Unknown | 405 | 263 | 156 | 129 |  | 953
    Primary Care Participants: number analyzed (Participants) | 70223 | 33650 | 46878 | 31291 | 0 | 182042
    Primary Care Participants: White | 59513 | 17456 | 24280 | 14456 |  | 115705
    Primary Care Participants: Non-White | 4195 | 14620 | 20842 | 15203 |  | 54860
    Primary Care Participants: Unknown | 6515 | 1574 | 1756 | 1632 |  | 11477
    Staff: number analyzed (Participants) | 0 | 0 | 0 | 0 | 27 | 27
    Staff: White |  |  |  |  | 25 | 25
    Staff: Non-White |  |  |  |  | 2 | 2
    Staff: Unknown |  |  |  |  | 0 | 0
Sleep Medication [Count of Participants; unit: Participants] — Participants from all sites identified in the Implementation phase in PCMHI and Primary Care, and Staff from all sites identified among all phases. Population: Staff - sleep medication not measured
  Participants
    PCMHI Participants: number analyzed (Participants) | 4924 | 3927 | 2975 | 2258 | 0 | 14084
    PCMHI Participants: Yes | 556 | 243 | 452 | 138 | 0 | 1389
    PCMHI Participants: No | 4368 | 3684 | 2523 | 2120 | 0 | 12695
    Primary Care Participants: number analyzed (Participants) | 70223 | 33650 | 46878 | 31291 | 0 | 182042
    Primary Care Participants: Yes | 4483 | 1404 | 4094 | 1027 |  | 11008
    Primary Care Participants: No | 65740 | 32246 | 42784 | 30264 |  | 171034

OUTCOME MEASURES:

1. Primary Outcome: Veteran Participants Who Engaged in BBTI
Description: The number of Veterans in PCMHI who engaged in BBTI as indicated in the medical records
Time Frame: 54 months; All study phases (pre-training; pre-implementation; implementation; post-implementation)
Population: Veterans in PCMHI who engaged in BBTI
Measure: Count of Participants; unit: Participants
Arm/Group | Minneapolis VAMC | Philadelphia VAMC | Durham VAMC | Baltimore VAMC
Number analyzed (Participants) | 434 | 78 | 361 | 192
Participants
  Pre-Training | 14 | 1 | 21 | 0
  Pre-Implementation | 0 | 14 | 90 | 67
  Implementation | 203 | 35 | 88 | 50
  Post-Implementation | 217 | 28 | 162 | 75
Statistical Analysis 1: Comparison: Minneapolis VAMC; pre-training to implementation; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 15.61, 95% CI 2-sided [8.99 to 21.11]
Statistical Analysis 2: Comparison: Philadelphia VAMC; pre-implementation to implementation; Test type: Superiority; p = 0.18, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.81 to 3.00]
Statistical Analysis 3: Comparison: Durham VAMC; pre-implementation to implementation; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.17 to 2.22]
Statistical Analysis 4: Comparison: Baltimore VAMC; pre-implementation to implementation; Test type: Superiority; p = 0.48, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.77 to 1.76]

2. Secondary Outcome: Veterans in PCMHI Identified With Insomnia
Description: The number of Veterans with encounters in PCMHI related to insomnia, indicated by an insomnia diagnostic code and/or insomnia-related medication.
Time Frame: 54 months; All study phases (pre-training; pre-implementation; implementation; post-implementation)
Measure: Count of Participants; unit: Participants
Arm/Group | Minneapolis VAMC | Philadelphia VAMC | Durham VAMC | Baltimore VAMC
Number analyzed (Participants) | 2255 | 924 | 2386 | 1141
Participants
  Pre-Training | 718 | 314 | 717 | 354
  Pre-Implementation | 0 | 167 | 778 | 327
  Implementation | 857 | 280 | 505 | 217
  Post-Implementation | 680 | 163 | 386 | 243

3. Secondary Outcome: Veterans in Primary Care Identified With Insomnia
Description: The number of Veterans with encounters in Primary Care related to insomnia, indicated by an insomnia diagnostic code and/or insomnia-related medication.
Time Frame: 54 months; All study phases (pre-training; pre-implementation; implementation; post-implementation)
Measure: Count of Participants; unit: Participants
Arm/Group | Minneapolis VAMC | Philadelphia VAMC | Durham VAMC | Baltimore VAMC
Number analyzed (Participants) | 17693 | 8728 | 23757 | 7799
Participants
  Pre-Training | 6383 | 2737 | 7038 | 2378
  Pre-Implementation | 0 | 1875 | 6547 | 2383
  Implementation | 6135 | 2257 | 5482 | 1571
  Post-Implementation | 5175 | 1859 | 4690 | 1467

4. Secondary Outcome: BBTI Effectiveness (Intent to Treat)
Description: Change on the Insomnia Severity Index (ISI; 0-28, low scores indicate lower severity) from the initial score obtained (e.g., PCMHI initial evaluation, BBTI session 1) to the final score documented in medical records. Data aggregated across phases (averaged) for first session and last session.
Time Frame: 42 months; during the pre-implementation, implementation, and post-implementation phases. Time from BBTI first session to BBTI last session varies, but can range 1-13 weeks.
Population: This is the intent to treat (ITT) analysis and all ISI data are included from participants who initiated BBTI. Results provided for all sites combined and individual sites. Data at the participant-level (Veterans in PCMHI), with data extracted from BBTI progress notes in the electronic health records, retrospectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BBTI First Session: Insomnia Severity Index (ISI) obtained from BBTI first session documented in progress notes and extracted from the electronic medical records.
- BBTI Last Session: Insomnia Severity Index (ISI) obtained from BBTI last session documented in progress notes and extracted from the electronic medical records.
Arm/Group | BBTI First Session | BBTI Last Session
Number analyzed (Participants) | 515 | 183
score on a scale
  All Sites | 16.85 (5.79) | 13.41 (7.02)
  Minneapolis VAMC: number analyzed (Participants) | 229 | 52
  Minneapolis VAMC | 16.09 (5.46) | 11.40 (7.60)
  Philadelphia VAMC: number analyzed (Participants) | 63 | 35
  Philadelphia VAMC | 18.30 (5.32) | 13.69 (6.17)
  Durham VAMC: number analyzed (Participants) | 153 | 69
  Durham VAMC | 18.05 (6.03) | 14.30 (6.69)
  Baltimore VAMC: number analyzed (Participants) | 70 | 27
  Baltimore VAMC | 18.36 (5.34) | 12.70 (6.99)
Statistical Analysis 1: Comparison: BBTI First Session vs BBTI Last Session; Test type: Superiority; p < 0.0001, Mixed Models Analysis; effect size for mixed effects model = 0.72
Statistical Analysis 2: Comparison: BBTI First Session vs BBTI Last Session; Minneapolis VAMC; Test type: Superiority; p < 0.0001, Mixed Models Analysis; effect size for mixed effects model = 0.83
Statistical Analysis 3: Comparison: BBTI First Session vs BBTI Last Session; Philadelphia VAMC; Test type: Superiority; p < 0.0001, Mixed Models Analysis; effect size for mixed effects model = 0.79
Statistical Analysis 4: Comparison: BBTI First Session vs BBTI Last Session; Durham VAMC; Test type: Superiority; p < 0.0001, Mixed Models Analysis; effect size for mixed effects model = 0.60
Statistical Analysis 5: Comparison: BBTI First Session vs BBTI Last Session; Baltimore VAMC; Test type: Superiority; p < 0.0001, Mixed Models Analysis; effect size for mixed effects model = 1.01

5. Secondary Outcome: BBTI Effectiveness (Per Protocol)
Description: as for outcome 4
Time Frame: 42 months; during the pre-implementation, implementation, and post-implementation phases. Time from BBTI first session to BBTI last session varies, but can range 2-13 weeks.
Population: This is the per protocol (PP) analysis and all ISI data are included from participants who completed at least 3 sessions of BBTI. Results provided for all sites combined and individual sites. Data at the participant-level (Veterans in PCMHI), with data extracted from BBTI progress notes in the electronic health records, retrospectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BBTI First Session: Insomnia Severity Index (ISI) from the initial score obtained from BBTI first session.
- BBTI Last Session: Insomnia Severity Index (ISI) from the initial score obtained from BBTI last session.
Arm/Group | BBTI First Session | BBTI Last Session
Number analyzed (Participants) | 101 | 101
score on a scale
  All Sites | 18.48 (5.42) | 12.31 (6.38)
  Minneapolis VAMC: number analyzed (Participants) | 16 | 16
  Minneapolis VAMC | 17.13 (4.70) | 8.13 (6.04)
  Philadelphia VAMC: number analyzed (Participants) | 24 | 24
  Philadelphia VAMC | 18.88 (5.34) | 13.79 (5.84)
  Durham VAMC: number analyzed (Participants) | 41 | 41
  Durham VAMC | 18.00 (6.14) | 13.00 (6.19)
  Baltimore VAMC: number analyzed (Participants) | 20 | 20
  Baltimore VAMC | 20.05 (4.32) | 12.45 (6.71)
Statistical Analysis 1: Comparison: BBTI First Session vs BBTI Last Session; All Sites; Test type: Superiority; p < 0.0001, Mixed Models Analysis; effect size for mixed effects model = 1.05
Statistical Analysis 2: Comparison: BBTI First Session vs BBTI Last Session; Minneapolis VAMC; Test type: Superiority; p < 0.0001, Mixed Models Analysis; effect size for mixed effects model = 1.72
Statistical Analysis 3: Comparison: BBTI First Session vs BBTI Last Session; Philadelphia VAMC; Test type: Superiority; p < 0.0001, Mixed Models Analysis; effect size for mixed effects model = 0.93
Statistical Analysis 4: Comparison: BBTI First Session vs BBTI Last Session; Durham VAMC; Test type: Superiority; p < 0.0001, Mixed Models Analysis; effect size for mixed effects model = 0.82
Statistical Analysis 5: Comparison: BBTI First Session vs BBTI Last Session; Baltimore VAMC; Test type: Superiority; p < 0.0001, Mixed Models Analysis; effect size for mixed effects model = 1.38

6. Secondary Outcome: PCMHI Providers (Staff) Who Delivered (Adopted) BBTI
Description: PCMHI providers (Staff) who delivered (adopted) BBTI (adopted) to at least 1 Veteran - measured in each phase (pre-implementation, implementation, post-implementation).
Time Frame: 42 months; during the pre-implementation, implementation, and post-implementation phases.
Population: Number of PCMHI providers who delivered BBTI relative to providers who were eligible to deliver BBTI. Not all of these providers were considered enrolled in the study.
Measure: Number; unit: providers
Groups:
- Minneapolis VAMC: All sites underwent a 12-month pre-training period (phase 1) before undergoing training (month 0) for BBTI. Then sites were randomized to 0, 6, 12, or 18 months of the Pre-Implementation (phase 2), followed by 12 months of Implementation (phase 3, ERIC strategies were accessible and supported during this phase), and 12 months of Post-Implementation monitoring (phase 4).
  *This site was assigned to: Pre-Training, then Implementation (Month 1 - Month 12), then Post-Implementation (Month 13-24). Note, this site was randomized to skip Pre-Implementation (phase 2).
  **Data includes Implementation and Post-Implementation.
- Philadelphia VAMC: All sites underwent a 12-month pre-training period (phase 1) before undergoing training (month 0) for BBTI. Then sites were randomized to 0, 6, 12, or 18 months of the Pre-Implementation (phase 2), followed by 12 months of Implementation (phase 3, ERIC strategies were accessible and supported during this phase), and 12 months of Post-Implementation monitoring (phase 4).
  *This site was assigned to: Pre-Training, then Pre-Implementation (Month 1-6), Implementation (Month 7-18), then Post-Implementation (Month 19-30).
  **Data includes Pre-Implementation, Implementation and Post-Implementation.
- Durham VAMC: All sites underwent a 12-month pre-training period (phase 1) before undergoing training (month 0) for BBTI. Then sites were randomized to 0, 6, 12, or 18 months of the Pre-Implementation (phase 2), followed by 12 months of Implementation (phase 3, ERIC strategies were accessible and supported during this phase), and 12 months of Post-Implementation monitoring (phase 4).
  *This site was assigned to: Pre-Training, then Pre-Implementation (Month 1-12), Implementation (Month 13-24), then Post-Implementation (Month 25-36).
  **Data includes Pre-Implementation, Implementation and Post-Implementation.
- Baltimore VAMC: All sites underwent a 12-month pre-training period (phase 1) before undergoing training (month 0) for BBTI. Then sites were randomized to 0, 6, 12, or 18 months of the Pre-Implementation (phase 2), followed by 12 months of Implementation (phase 3, ERIC strategies were accessible and supported during this phase), and 12 months of Post-Implementation monitoring (phase 4).
  *This site was assigned to: Pre-Training, then Pre-Implementation (Month 1-18), Implementation (Month 19-30), then Post-Implementation (Month 31-42).
  **Data includes Pre-Implementation, Implementation and Post-Implementation.
Arm/Group | Minneapolis VAMC | Philadelphia VAMC | Durham VAMC | Baltimore VAMC
Number analyzed (Participants) | 91 | 142 | 94 | 82
providers
  Pre-Implementation: number analyzed (Participants) | 0 | 142 | 94 | 82
  Pre-Implementation |  | 17 | 33 | 17
  Implementation | 23 | 29 | 27 | 17
  Post-Implementation | 27 | 20 | 27 | 17

7. Secondary Outcome: Implementation/Treatment Fidelity (Staff)
Description: Mean Competency Rating Score (0-36, higher scores indicate higher competency, >17 indicates competency)
  PCMHI providers (Staff) were measured via mock treatment sessions by site PIs/subject matter experts using the BBTI-Competency Rating Scale (BBTI-CRS) during the pre-implementation, implementation, and post-implementation phases. Overall refers to aggregate ratings (averaged) from all phases in which BBTI-CRS was delivered - providers could complete up to 5 ratings (up to 3 for pre-implementation, 1 for implementation, and 1 for post-implementation).
Time Frame: 42 months; the BBTI-CRS was administered during pre-implementation (up to 3 times), implementation (1 time, at the end), and post-implementation (1 time, at the end)
Population: PCMHI providers (Staff) trained in BBTI who consented to participate in the competency ratings. Not all Staff completed ratings at all phases and there was no plan to compare between sites. Only descriptive statistics (Mean/Standard Deviation) reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BBTI Competency: PCMHI clinicians who were rated using the BBTI-CRS by Site PIs/subject matter experts.
Arm/Group | BBTI Competency
Number analyzed (Participants) | 18
score on a scale
  Overall (phases 2-4) | 31.46 (5.14)
  Pre-Implementation (phase 2) | 31.02 (5.57)
  Implementation (phase 3): number analyzed (Participants) | 14
  Implementation (phase 3) | 33.64 (3.52)
  Post-Implementation (phase 4): number analyzed (Participants) | 11
  Post-Implementation (phase 4) | 33.55 (2.77)

8. Secondary Outcome: Barriers & Facilitators (CFIR Determinants)
Description: Strength and valence rating for identified barriers and facilitators (determinants) from the Consolidated Framework for Implementation Research (CFIR) qualitative interviews. CFIR determinants, identified through qualitative interviews with PCMHI providers, were rated on strength (0, 1, 2; higher numbers indicate stronger influence) and valence (- indicates negative/harmful influence; + indicates positive/helpful influence) to determine how helpful or harmful an identified CFIR determinant is for implementing BBTI in PCMHI. Ratings were aggregated across sites and phases (consensus by 3 raters with adjudication by PI as needed).
Time Frame: 42 months; qualitative interviews took place at the end of the pre-implementation, implementation, and post-implementation phases.
Population: 16 Staff participants were engaged in CFIR interviews with 3 study team members coding the interviews and conducting strength and valence ratings. Strength (0, 1, 2) and valence (- / +) ratings help to determine how helpful or harmful an identified CFIR determinant is for implementation of BBTI.
Measure: Number; unit: rating score for each CFIR determinant
Groups:
- Implementation Strategies: Implementation strategies aggregated from PCMHI providers (Staff) at all sites across the pre-implementation, implementation, and post-implementation phases.
Arm/Group | Implementation Strategies
Number analyzed (Participants) | 16
rating score for each CFIR determinant
  Innovation: Adaptability: number analyzed (Participants) | 3
  Innovation: Adaptability | 1
  Innovation: Trialability: number analyzed (Participants) | 3
  Innovation: Trialability | 1
  Innovation: Relative Advantage: number analyzed (Participants) | 3
  Innovation: Relative Advantage | 2
  Innovation: Design: number analyzed (Participants) | 3
  Innovation: Design | 2
  Outer: Partnerships & Connections: number analyzed (Participants) | 3
  Outer: Partnerships & Connections | 1
  Inner: Work Infrastructure: number analyzed (Participants) | 3
  Inner: Work Infrastructure | -2
  Inner: Communications: number analyzed (Participants) | 3
  Inner: Communications | 1
  Inner: Compatibility: number analyzed (Participants) | 3
  Inner: Compatibility | 2
  Inner: Mission Alignment: number analyzed (Participants) | 3
  Inner: Mission Alignment | 2
  Inner: Available Resources: number analyzed (Participants) | 3
  Inner: Available Resources | 1
  Inner: Access to Knowledge & Information: number analyzed (Participants) | 3
  Inner: Access to Knowledge & Information | 2
  Inner: Relative Priority: number analyzed (Participants) | 3
  Inner: Relative Priority | -1
  Individuals: Innovation Deliverers - Capability: number analyzed (Participants) | 3
  Individuals: Innovation Deliverers - Capability | 2
  Individuals: Innovation Recipients - Need: number analyzed (Participants) | 3
  Individuals: Innovation Recipients - Need | 2
  Individuals: Innovation Recipients - Motivation: number analyzed (Participants) | 3
  Individuals: Innovation Recipients - Motivation | -1
  Process: Teaming: number analyzed (Participants) | 3
  Process: Teaming | 2
  Process: Tailoring Strategies: number analyzed (Participants) | 3
  Process: Tailoring Strategies | 2
  Process: Engaging Recipients: number analyzed (Participants) | 3
  Process: Engaging Recipients | -1
  Process: Adapting: number analyzed (Participants) | 3
  Process: Adapting | 2

9. Secondary Outcome: Implementation Strategy Utilization Survey
Description: Indication of implementation strategy utilization (yes/no) and rating of its importance (1 = not at all important, 5 = very important) and feasibility ((1 = not at all feasible, 5 = very feasible).
Time Frame: 12 months: 4 times - every 3-months during the Implementation phase.
Population: This measure was abandoned during the study, early on with no data collected, since much of the data intended to be collected through this survey could be captured/collected as part of the CFIR interviews and ratings (Outcome #8).
Groups:
- Implementation Strategy Utilization Survey: Indication of implementation strategy utilization (yes/no) and rating of its importance (1 = not at all important, 5 = very important) and feasibility ((1 = not at all feasible, 5 = very feasible).
Arm/Group | Implementation Strategy Utilization Survey
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Not Applicable; Deaths and Adverse Events were not monitored/assessed for Veteran Participants nor Staff
Description: Not Applicable; Deaths and Adverse Events were not monitored/assessed for Veteran Participants nor Staff
Groups:
- EG000: Not Applicable; Deaths and Adverse Events were not monitored/assessed for Veteran Participants nor Staff
Arm/Group | EG000
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT04350866/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT04350866/ICF_002.pdf